CLINICAL TRIAL: NCT00911404
Title: Comparison of Two Different Diets Containing Different Proportions of Carbohydrates in the Treatment of Gestational Diabetes Mellitus: A Randomized Clinical Trial
Brief Title: Carbohydrate Restriction for Gestational Diabetes Mellitus
Acronym: LO-CA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Arnau de Vilanova (Other)
Responsible Party: Principal Investigator, Marta Hernández García, MD, Hospital Arnau de Vilanova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIC-670
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: Gestational diabetes; Carbohydrate; Diet; Insulin
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low CHO (Experimental): Diet with 40% total calories from carbohydrates.
  Interventions: Behavioral: Low CHO
- High CHO (Active Comparator): Diet with 55% total calories from carbohydrates.
  Interventions: Dietary Supplement: High CHO diet

INTERVENTIONS:
Behavioral: Low CHO — Diet with 40% total calories from carbohydrates. In the "Low-CHO" arm, 15% of calories from carbohydrates will be substituted by monounsaturated fat.
  Arms: Low CHO
Dietary Supplement: High CHO diet — Diet with 55% total calories from carbohydrates.
  Arms: High CHO

SUMMARY:
There is evidence that controlling total amount of carbohydrates is a strategy for controlling glucose levels in diabetes mellitus. There is not major evidence that any given macronutrient percentage may be recommended to treat a woman with Gestational Diabetes Mellitus (GDM). In the investigators' country, insulin is the second-line treatment once medical nutrition therapy (MNT) has failed to control glucose levels during pregnancy. Insulin treatment is more expensive and not as well accepted as MNT. The investigators have designed a randomized-controlled trial to assess whether a diet with 40% total calories from carbohydrates may reduce the need of insulin treatment in women with gestational diabetes, without having unfavourable pregnancy outcomes, in comparison with a diet with 55% total calories from carbohydrates.

ELIGIBILITY:
Inclusion Criteria:

* Gestational diabetes mellitus
* Single pregnancy

Exclusion Criteria:

* Multiple pregnancy
* High risk pregnancy (any other concomitant illness, excluding hypertension and obesity)
* Low ability to understand and follow a diet
* Need to use insulin different from regular insulin

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2009-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Need of insulin treatment for GDM | Day of delivery

SECONDARY OUTCOMES:
Time from GDM diagnosis free of insulin treatment | Day of delivery
Maternal ketonemia and/or ketonuria | Day of delivery
Maternal morbidity | Day of delivery
Fetal morbidity | 1 month after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Didac Mauricio, MD PhD, Study Director — Hospital Universitari Arnau de Vilanova; Marta Hernández, MD, Principal Investigator — Hospital Universitari Arnau de Vilanova
Locations (1):
- Hospital Universitari Arnau de Vilanova, Lleida, Lleida, Spain

REFERENCES:
- [Background] Cypryk K, Kaminska P, Kosinski M, Pertynska-Marczewska M, Lewinski A. A comparison of the effectiveness, tolerability and safety of high and low carbohydrate diets in women with gestational diabetes. Endokrynol Pol. 2007 Jul-Aug;58(4):314-9. PMID 18058723
- [Background] Peterson CM, Jovanovic-Peterson L. Percentage of carbohydrate and glycemic response to breakfast, lunch, and dinner in women with gestational diabetes. Diabetes. 1991 Dec;40 Suppl 2:172-4. doi: 10.2337/diab.40.2.s172. PMID 1748252
- [Background] Major CA, Henry MJ, De Veciana M, Morgan MA. The effects of carbohydrate restriction in patients with diet-controlled gestational diabetes. Obstet Gynecol. 1998 Apr;91(4):600-4. doi: 10.1016/s0029-7844(98)00003-9. PMID 9540949
- [Derived] Moreno-Castilla C, Hernandez M, Bergua M, Alvarez MC, Arce MA, Rodriguez K, Martinez-Alonso M, Iglesias M, Mateu M, Santos MD, Pacheco LR, Blasco Y, Martin E, Balsells N, Aranda N, Mauricio D. Low-carbohydrate diet for the treatment of gestational diabetes mellitus: a randomized controlled trial. Diabetes Care. 2013 Aug;36(8):2233-8. doi: 10.2337/dc12-2714. Epub 2013 Apr 5. PMID 23564917